CLINICAL TRIAL: NCT00000766
Title: CMV Retinitis Retreatment Trial
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Purpose: Treatment
Other Study IDs: ACTG 228
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2011-03-01 (Estimated); Status verified 2011-02

CONDITIONS: Cytomegalovirus Retinitis; HIV Infections
Keywords: Retinitis; Ganciclovir; Foscarnet; Cytomegalovirus Infections; Acquired Immunodeficiency Syndrome
MeSH Terms: conditions — Cytomegalovirus Retinitis; HIV Infections; Retinitis; Multiple Acyl Coenzyme A Dehydrogenase Deficiency; Cytomegalovirus Infections; Acquired Immunodeficiency Syndrome | interventions — Foscarnet; Ganciclovir

INTERVENTIONS:
Drug: Foscarnet sodium
Drug: Ganciclovir

SUMMARY:
To assess the safety and efficacy of three therapeutic regimens (foscarnet, ganciclovir, or the combination) for recurrent or persistent AIDS-related cytomegalovirus (CMV) retinitis.

Although therapy with foscarnet or ganciclovir halts retinitis progression in 90 percent of patients treated, relapses are common and may accelerate due to development of drug resistance, deteriorating immune function, or other factors. Treatment strategies currently being investigated include switching patients from one drug to the other or combining the two drugs.

DETAILED DESCRIPTION:
Although therapy with foscarnet or ganciclovir halts retinitis progression in 90 percent of patients treated, relapses are common and may accelerate due to development of drug resistance, deteriorating immune function, or other factors. Treatment strategies currently being investigated include switching patients from one drug to the other or combining the two drugs.

Patients are randomized to receive foscarnet, ganciclovir, or a combination of the two drugs (administered sequentially). Initially, patients undergo single or multiple cycles of induction therapy for 14 days followed by maintenance therapy. Patients in whom the retinitis continues to progress or who are intolerant of the initial treatment switch to the alternative drug for further cycles of induction and maintenance. Patients on the combination arm in whom retinitis continues to progress are given further cycles of the combination at an increased dose, or, if one drug is causing toxicity, are given further cycles with the alternative drug. Patients are followed monthly for 6 months and then every 3 months thereafter.

ELIGIBILITY:
Inclusion Criteria

Required:

* At least 28 days of prior foscarnet or ganciclovir.

Concurrent Medication:

Allowed:

* G-CSF.

Recommended:

* Antiretroviral therapy.

Patients must have:

* HIV infection or AIDS.
* Active CMV retinitis after 28 or more days of either foscarnet or ganciclovir therapy.
* At least one lesion with one-quarter disk area or more that can be photographed.
* Visual acuity of 3 or more letters on ETDRS chart (5/200 Snellen) in an affected eye.

Exclusion Criteria

Co-existing Condition:

Patients with the following symptoms and conditions are excluded:

* Media opacity severe enough to preclude visualization of both fundi.
* Retinal detachment not scheduled for surgical repair.

Patients with the following prior conditions are excluded:

* History of intolerance to ganciclovir or foscarnet sufficient to contraindicate use.
* History of combination foscarnet/ganciclovir therapy.

Active drug or alcohol abuse sufficient to prevent compliance.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300
Dates: Primary Completion 1995-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (9):
- United States (9):
  - UCSD - Shiley Eye Ctr / SOCA, La Jolla, California
  - UCLA - Jules Stein Eye Institute / SOCA, Los Angeles, California
  - UCSF - San Francisco Gen Hosp, San Francisco, California
  - Northwestern Univ / SOCA, Chicago, Illinois
  - Johns Hopkins Hosp / SOCA, Baltimore, Maryland
  - New York Univ Med Ctr / SOCA, New York, New York
  - New York Hosp - Cornell Med Ctr / Sloan - Kettering / SOCA, New York, New York
  - Mount Sinai Med Ctr / SOCA, New York, New York
  - Univ of North Carolina / SOCA, Chapel Hill, North Carolina

REFERENCES:
- [Background] Jabs DA. Design of clinical trials for drug combinations: cytomegalovirus retinitis--foscarnet and ganciclovir. The CMV retinitis retreatment trial. Antiviral Res. 1996 Jan;29(1):69-71. doi: 10.1016/0166-3542(95)00921-3. PMID 8721550